CLINICAL TRIAL: NCT00223041
Title: Cardiovascular Events in Renal Transplant Recipients With Low LDL-cholesterol Receiving Tacrolimus in Combination With the Statin Fluvastatin
Brief Title: Cranoc Lipid Study in Renal Transplantation
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No possibilty to receive all plened patients for this study
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: L. Renders, University of Kiel, department of Nephrology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2006-05

CONDITIONS: Renal Transplantation
Keywords: renal transplantation; cardiovasculary disease; statin
MeSH Terms: interventions — Fluvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (therapy with fluvastatin 80mg retard) (No Intervention): kidney transplants receive in addition fluvastatin 80mg retard for 3 years
- B (Placebo Comparator): no therapy with fluvastatin
  Interventions: Drug: Fluvastatin

INTERVENTIONS:
Drug: Fluvastatin — Arm A receives fluvastatin Arm b receives no fluvastatin
  Arms: B

SUMMARY:
Cardiovascular disease after renal transplantation is an important problem. Patients after renal transplantation with low LDL-Levels (<130mg/dl) receive Fluvastatin 80mg/day (or no medication, to look for the cardiovascular outcome with and without statins.

DETAILED DESCRIPTION:
Cardiovascular disease after renal transplantation is an important problem. Patients after renal transplantation with low LDL-Levels (<130mg/dl) receive Fluvastatin 80mg/day (or no medication, to look for the cardiovascular outcome with and without statins.

ELIGIBILITY:
Inclusion Criteria:

* patients (18 - 65, inclusive)
* cadaver and living kidney transplantation (1. Ntx, 2. Ntx)
* LDL-cholesterol ≤ 130mg/dl (-3 Mo until start of Tx)
* Patients with a history of Myocard infarct: LDL-Cholesterol ≤ 110mg/dl
* Immunsuppression: Tacrolimus in combination with steroids or Mycophenolat Mofetil
* patients indulgence

Exclusion Criteria:

* statin before the study

  * LDL-Cholesterol >130mg/dl before transplantation
  * Instabil Angina, Myocard infarct <6 months before transplantation
  * symptomatic Hypothyreosis
  * child bearing, lactating
  * elavated liver encymes (> 2x elavated: AST, ALT, bilirubine, PCK)
  * Fibrates are not allowed
  * multiorgantransplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2003-04; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
cardivasculary events (cardiovaskulary, cerebrovaskulary, peripher vaskulary) | during the study

SECONDARY OUTCOMES:
patients and kidney survival | during the study
amount and typ of rejection (Banff-classifikation) | during the study
change in lipids | during the study
adverse events of the statin fluvastatin | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Renders, MD, Principal Investigator — University of Scghleswig-Holstein, Campus Kiel, Department of Nephrology
Locations (1):
- University of Schleswig-Holstein, Campus Kiel, Department of Nephrology, Kiel, Germany